CLINICAL TRIAL: NCT06924502
Title: Non-controlled, Exploratory, Single-arm Clinical Study With a Water-in-oil Emulsion to Test the Protecting and Caring Effect of the Formulation on 'Incontinence-care Product Requiring' Fecal and/or Urinary Incontinent Patients
Brief Title: Testing the Protective and Caring Effect of a Water-in-oil Formulation in Patients Suffering From Urinary and/or Fecal Incontinence and Requiring Incontinence Care Products
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLS-02/2024
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Incontinence, Urinary; Incontinence, Fecal
MeSH Terms: conditions — Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Masking Description: Blinding of sponsor label (blanco primary packaging)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test Product (P-001230/2) (Experimental): Patients receive at least two applications of the test product P-001230/2 in the application area every day. An additional washing product is used to clean the skin.
  Interventions: Other: Protective Balm

INTERVENTIONS:
Other: Protective Balm — The test product will be applied in addition to an additional washing product in the test area.

SUMMARY:
The aim of this study is to test the protecting and caring effect of a protective balm on patients suffering from urinary and/or fecal incontinence and need incontinence care products.

DETAILED DESCRIPTION:
Patients receive at least two applications of the test product in the application area daily for two weeks. An additional washing product is used during the entire application time. The caring and skin protecting effects, the skin tolerability and cosmetic efficacy of the test product will be assessed by a physician, a nurse and the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient is capable of understanding the information given to them and providing informed consent
* 70 years of age and older
* Patients with incontinence (fecal and/or urinary), requiring incontinence protection material
* Skin type on Fitzpatrick scale: Between I to IV

Exclusion Criteria:

* Current cancer treatment such as chemotherapy, irradiation
* Documented allergies to skin care and / or skin cleansing products
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, etc. at the test area that could influence the investigation
* Incontinence-associated dermatitis (IAD) stage >1a
* Active skin disease at the test area
* Any topical medication at the test area within the last 3 days prior to the start of the study and / or hroughout te entire course of the study
* Mini-Mental-Status-Test (MMST) < 20

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of skin tolerability (single parameters) by the physician regarding erythema, oedema, dryness, papules or pustules | Day 1 vs Day 15±2 (after 2 weeks of test product application)
  Single parameters (erythema, oedema, dryness, papules or pustules) will be assessed by a scale.
Global assessment of tolerability by the phyisician | Day 15 ±2 (after 2 weeks of test product application)
  The physician will evaluate the global skin tolerability, according to a scale (taking results of skin tolerability (single parameters), and his or her personal assessment of tolerability at all time points into account).
Global assessment of cosmetic efficacy by the physician | Day 15 ±2 (after 2 weeks of test product application)
  The physician will evaluate the global efficacy, according to a scale.
Assessment of skin condition by a nurse | Day 1 and Day 15 ±2 (after 2 weeks of test product application)
  The skin condition (color, turgor and surface of the skin) will be assessed by binary queries (yes/no).
  The caring and protecting status of the skin will be assessed by an Visual Analogue Scale (VAS).
Assessment of product characteristics by a nurse | Day 15 ±2 (after 2 weeks of test product application)
  Product characteristics regarding scent, spreadability, removability, appearance of the skin (redness, dryness) will be assessed by a questionnaire with predefined answer options.
Global assessment of the product by a nurse | Day 15 ±2 (after 2 weeks of test product application)
  The nurse will evaluate the global assessment of the product, according to a scale (taking results of the skin condition regarding the caring and protecting status and the product characteristics into account).
Assessment of product characteristics | Day 15 ±2 (after 2 weeks of test product application)
  Product characteristics will be assessed by the patient in a questionnaire regarding sensation during application of the product by the nurse (feeling during application on the skin).
Assessment of skin tolerability by the patient | Day 15 ±2 (after 2 weeks of test product application)
  The overall subjective skin status after application of the test product will be evaluated summarized for the whole application period according to a scale (each parameter (itching, burning, stinging, pain, soreness) separately).

OTHER OUTCOMES:
Assessment of urine incontinence | Day 1
  Assessment of urine incontinence according to ICIQ-SF questionnaire.
Assessment of fecal incontinence | Day 1
  Assessment of fecal incontinence according to CCFIS questionnaire.
Product use | Day 15 ±2 (after 2 weeks of test product application)
  Product is weighed before and after the application period

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Dortmund, Dortmund, Germany